CLINICAL TRIAL: NCT01334645
Title: Diagnostic Value of Copeptin Assay for Acute Coronary Syndrome Without ST-segment Elevation
Brief Title: Copeptin and Acute Coronary Syndrome Without ST-segment Elevation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Collaborators: Association des Médecins des Urgences de Clermont-Ferrand (Other); BRAHMS Biomarkers (Unknown); General Hospital Henri Mondor, Aurillac, France (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Diagnostic
Other Study IDs: CHU-0092; 2010-A01186-33
Record Dates: First submitted 2011-04-11; First posted 2011-04-13 (Estimated); Last update posted 2013-05-29 (Estimated); Status verified 2013-05

CONDITIONS: Chest Pain
Keywords: Copeptin; Troponin; Diagnosis; Chest pain; Acute Coronary Syndrome; Acute Myocardial Infarction; Unstable Angina
MeSH Terms: conditions — Chest Pain; Diabetes Insipidus; Disease; Acute Coronary Syndrome; Angina, Unstable | interventions — Arginine Vasopressin

STUDY DESIGN:
Who Masked: Participant

INTERVENTIONS:
Other: Copeptin — Patients with hyponatremia < 135 mmol/L or troponin > 1 μg/L are released study.
  Blood sampling are taken for Troponine T, myoglobin, creatin kinase and copeptine analysis and 18-lead ECG was performed after 2, 4, 6 and 12 h.
  Copeptin and myoglobin are measured at the end of the patients inclusion, after to be centrifugrd end frozen at -80°C at each time point.
  The treatment of patients is not modified by the study. At 90 days, clinicals and paraclinicals events are collected

SUMMARY:
The purpose of this study is to determine whether the combination of copeptine and troponin adds diagnosis information to that provided by troponin alone or the combination of troponin and myoglobin.

Hypothesis : If the values of troponin and copeptin are not elevated, diagnosis of acute myocardial infarction can be ruled out without prolonged monitoring and serial blood sampling.

DETAILED DESCRIPTION:
Patients older than 18 years with pain suggestive of Acute Coronary Syndrome, with onset within the last 12 hours, presenting to the Emergency Department of the University Hospital Gabriel Montpied (Clermont-Ferrand, France) and the General Hospital Henri Mondor (Aurillac, France) are enrolled.

Upon admission to the hospital, all patient underwent an initial clinical assessment, including medical history, temperature, respiratory rate, cardiac frequency, blood pressure, pulse oxymetry, 18-lead ECG, chest X-ray and screening blood test including C reactive protein, natremia, Troponine T, myoglobin, creatin kinase and copeptine.

Patients with hyponatremia < 135 mmol/L or troponin > 1 μg/L are released study.

Blood sampling are taken for Troponine T, myoglobin, creatin kinase and copeptine analysis and 18-lead ECG was performed after 2, 4, 6 and 12 h.

Copeptin and myoglobin are measured at the end of the patients inclusion, after to be centrifugrd end frozen at -80°C at each time point.

The treatment of patients is not modified by the study. At 90 days, clinicals and paraclinicals events are collected.

ELIGIBILITY:
Inclusion Criteria:

* Chest pain suggestive of Acute Coronary Syndrome
* Chest pain with onset within the last 12 h
* Patients older than 18 years

Exclusion Criteria:

* ST-Elevation Myocardial infarction
* Legal incapacity
* Sepsis
* Hyponatremia < 135 mmol/L
* Shock
* Lung neoplasms
* life expectancy of less than 6 months
* Refuse to consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 134 (Actual)
Dates: Start 2011-03; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Copeptin value | at day 1

SECONDARY OUTCOMES:
Troponin, Myoglobin and Creatin Kinase values. Clinicals and paraclinicals events . | at 90 days

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan DUCHENNE, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU Clermont-Ferrand, Clermont-Ferrand, France

REFERENCES:
- [Derived] Duchenne J, Mestres S, Dublanchet N, Combaret N, Marceau G, Caumon L, Dutoit L, Ughetto S, Motreff P, Sapin V, Schmidt J; NSTEMI Study. Diagnostic accuracy of copeptin sensitivity and specificity in patients with suspected non-ST-elevation myocardial infarction with troponin I below the 99th centile at presentation. BMJ Open. 2014 Mar 24;4(3):e004449. doi: 10.1136/bmjopen-2013-004449. PMID 24662448